CLINICAL TRIAL: NCT00331084
Title: Efficacy of Antibiotic Steroid Combination Compared With Individual Administration in Prevention of Postoperative Inflammation in Patients Having Cataract Surgery
Brief Title: Efficacy/Safety of Antibiotic Steroid Combination in Prevention of Postoperative Inflammation in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Rubens Belfort Jr, Head Professor of Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BRA-05-01
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Inflammation Following Cataract Surgery
Keywords: prevention of post inflammation in cataract surgery
MeSH Terms: interventions — Anti-Bacterial Agents; Moxifloxacin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antibiotic steroid drops/single vial (Experimental): efficacy of antibiotic steroid combination compared with individual administration in prevention of postoperative inflammation in patients having cataract surgery
  Interventions: Drug: antibiotic/steroid combination
- antibiotic steroids drops (Active Comparator): efficacy of antibiotic steroid combination compared with individual administration in prevention of postoperative inflammation in patients having cataract surgery
  Interventions: Drug: moxifloxacin / dexamethasone

INTERVENTIONS:
Drug: antibiotic/steroid combination — 1 gtt, 4x/day, 15 days
  Other Names: moxifloxacin / dexamethasone
  Arms: antibiotic steroid drops/single vial
Drug: moxifloxacin / dexamethasone — 1 gtt 4x/day, 15 days
  Arms: antibiotic steroids drops

SUMMARY:
efficacy of antibiotic steroid combination compared with individual administration in prevention of postoperative inflammation in patients having cataract surgery

DETAILED DESCRIPTION:
Study of 15 +-1 day, double-masked, randomized, two arms, parallel groups to confirm the efficacy of antibiotic steroid combination compared with individual administration in prevention of postoperative inflammation in patients having cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* patients having cataract surgery

Exclusion Criteria:

* Uncontrolled glaucoma or intraocular hypertension;
* Use of any ocular anti-infectious drugs or any topical or systemic ocular NSAIDs during the study but study drugs;
* A history of chronic or recurrent ocular inflammatory disease;
* Uncontrolled diabetes mellitus and diabetic retinopathy ;
* Patients with sight in a single eye;
* Iris atrophy in the eye to be operated;
* Pregnant or lactating women, or women of childbearing potential who are not using proper birth-control methods;
* Known or suspected allergy or hypersensitivity to any component of study medication;
* A history or any other evidence of severe systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
day 15 evaluation of anterior chamber | 15 days pos-op

SECONDARY OUTCOMES:
day 15 evaluation of ocular pain, physician´s follow-up impression of inflammatory reaction score | 15 days pos-op

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort Jr, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Dept of Opthalmology - Rua Botucatu 824, São Paulo, São Paulo, Brazil